CLINICAL TRIAL: NCT02837744
Title: Safety and Efficacy of Axiostat® Hemostatic Dressing on Radial Access After Percutaneous Procedure
Brief Title: Studying Hemostatic Effect of Axiostat® Dressing on Radial Access After Percutaneous Procedure
Acronym: AHD
Status: Completed | Type: Observational
Sponsor: Axio Biosolutions Pvt. Ltd. (Other)
Responsible Party: Sponsor
Other Study IDs: ABPL/002; U1111-1185-5780 (Other: World Health Organization); CTRI/2016/07/007115 (Registry Identifier: Clinical Trial Registry - India)
Record Dates: First submitted 2016-07-11; First posted 2016-07-20 (Estimated); Results first posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-02

CONDITIONS: Percutaneous Coronary Intervention; Angiography; Angioplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Axiostat®: Size: 3.5 cm X 3.5 cm
  Interventions: Device: Axiostat®

INTERVENTIONS:
Device: Axiostat® — Axiostat Chitosan Hemostatic dressing belongs to an advanced class of wound dressing that stops bleeding within few minutes of application by providing an active mechanical barrier.
  Other Names: Hemostatic Dressing

SUMMARY:
To evaluate Safety and Efficacy of Axiostat® hemostatic dressing in terms of time to achieve hemostasis, post application complication and comfort levels of patients.

DETAILED DESCRIPTION:
To evaluate Safety and Efficacy of Axiostat® hemostatic dressing in terms of time to achieve hemostasis, post application complication and comfort levels of patients who have undergone radial intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years.
2. Patient and/or patient's legal representative and/or impartial witness has/have been informed of the nature of the study and agrees to its provision and has provided written informed consent as approved by the Ethics Committee of the investigative site.
3. Iatrogenic puncture
4. Patient who want to undergo radial intervention.
5. All puncture size must be less than 2.5cm.

Exclusion Criteria:

1. Prior diagnosis of disease or medical condition affecting the ability of blood to clot (e.g., hemophilia.).
2. Patients with known sensitivity to chitosan (shellfish) used in this study.
3. Patients who, in the opinion of the Investigator, may not complete the study for any reason, e.g. Patient requiring Immediate suturing.
4. Patient is currently participating in an investigational drug or dressing study that has not yet completed its primary endpoint interferes with procedure and assessments in this trial.
5. Pregnant women.
6. Patients with hemorrhagic shock.
7. Patient having hemoglobin < 9 g/dl.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All eligible patients who came to the institution/hospital and provided informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Milan Chag, Dr., Principal Investigator — Care Institute of Medical Sciences
Locations (1):
- Care Institute of Medical Sciences,Nr. Shukan Mall, Off Science City Road,Sola, Ahmedabad, Gujarat, India

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Axiostat®
Started | 70
Completed | 70
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Axiostat®
Number analyzed (Participants) | 70
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Males and Females have been mentioned separately
  years
    Males: number analyzed (Participants) | 53
    Males | 55.94 (12.23)
    Females: number analyzed (Participants) | 17
    Females | 56.35 (9.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 53
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  India | 70
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 28.27 (6.29)
Baseline Blood Pressure [Mean (Standard Deviation); unit: mmHg]
  Systolic Blood Pressure | 136 (20)
  Diastolic Blood Pressure | 81 (13)
Haemoglobin [Mean (Standard Deviation); unit: g/dl] | 13.4 (1.37)
Prior History and Risk Factors [Count of Participants; unit: Participants] — Patients prior medical history was noted after enrollment Count of participants was noted for each parameter
  Participants
    Diabetes | 24
    Hypertension | 41
    Prior Percutaneous Coronary Intervention | 3
    Hyperlipidemia | 2
    Smoking | 2
    Prior Myocardial Infarction | 1
    Prior Coronary Artery Bypass Graft | 1
    Cardiogenic Shock | 1

OUTCOME MEASURES:

1. Primary Outcome: Time to Achieve Hemostasis
Description: Time to achieve hemostasis by observing the time at which blood oozing through or from periphery of the dressing stops.
  Unit of measurement is minutes.
Time Frame: 1 Day
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Axiostat®
Number analyzed (Participants) | 70
minutes | 5.43 (1.36)

2. Secondary Outcome: Quantity of Product Used
Description: Number of Axiostat® required to achieve hemostasis. Unit of measurement is number.
Time Frame: 1 Day
Measure: Number; unit: unit
Arm/Group | Axiostat®
Number analyzed (Participants) | 70
unit | 1

3. Secondary Outcome: Number of Patients With Re-bleeding
Description: Number of patients will be counted (unit of measurement is number/count of patients) with re-bleeding after removal of Axiostat
Time Frame: 1 Day
Measure: Count of Participants; unit: Participants
Arm/Group | Axiostat®
Number analyzed (Participants) | 70
Participants | 1

4. Secondary Outcome: Number of Participants With Allergy/Skin Irritation and Hematoma Formation
Description: 1. Observing occurrence of Allergy/Skin Irritation at the puncture site
  2. Observation of formation of Hematoma and/or any vascular complication after removal of Axiostat®.
  Mode of Measurement for both of the above outcomes is Visual Observation.
  Skin irritation/Allergy: Occurrence of redness at the puncture site was noted as skin irritation/allergy Hematoma: Hematoma formation at the puncture site. Hematoma was defined as presence of ecchymosis (the escape of blood into the tissues from ruptured blood vessels) at access site.
Time Frame: Upto 2 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Axiostat®
Number analyzed (Participants) | 70
Participants | 0

5. Secondary Outcome: Ease of Use of Product
Description: Level of ease of use of Axiostat was recorded. The ease of application and removal of Axiostat was rated as Excellent or Good or Fair or Poor by the Clinician / Operator Mode of Measurement is Verbal Inquiry.
Time Frame: Upto 2 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Axiostat®
Number analyzed (Participants) | 70
Participants
  Application: Excellent | 15
  Application: Good | 52
  Application: Fair | 3
  Removal: Excellent | 13
  Removal: Good | 57
  Removal: Fair | 0

6. Secondary Outcome: Patient Comfort Level
Description: Patients comfort level for use of dressing was recorded. The patient was required to rate the comfort level of use of dressing in terms of pain and swelling at the puncture site.
  It was assessed by verbal inquiry and visual observation.
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Axiostat®
Number analyzed (Participants) | 70
Participants
  No swelling & pain | 59
  Minor swelling & pain | 11
  Tolerable swelling & pain | 0
  Intolerable swelling & pain | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected till the patient was discharged.
Description: Any occurrence of adverse event was be recorded on the Adverse Event CRF. The number of patients at risk of adverse event is minimum as the product under evaluation is an approved product and so associated risks are less.
Arm/Group | Axiostat®
All-Cause Mortality (participants affected / at risk) | 0/70
Serious Adverse Events (participants affected / at risk) | 0/70
Other Adverse Events (participants affected / at risk) | 0/70

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-31): https://cdn.clinicaltrials.gov/large-docs/44/NCT02837744/Prot_SAP_000.pdf